CLINICAL TRIAL: NCT01804244
Title: An Open-label, Single-dose Study to Investigate the Pharmacokinetics and Safety of TMC278 After Oral Administration of TMC278 25 mg Tablet Under Fed Condition in Healthy Japanese Adult Male Subjects
Brief Title: A Single-Dose Pharmacokinetics and Safety Study of TMC278 in Healthy Adult Japanese Participants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR101181; TMC278IFD4005 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2013-03-01; First posted 2013-03-05 (Estimated); Last update posted 2014-03-19 (Estimated); Status verified 2014-03

CONDITIONS: Healthy
Keywords: Healthy; Pharmacokinetics; Japanese
MeSH Terms: interventions — Rilpivirine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TMC278 (Experimental): All participants will receive a single-dose of TMC278 (1 25-mg tablet [27.5 mg as the hydrochloride salt]) after an overnight fast (going without food) of at least 10 hours before eating a standard breakfast. Study drug will be taken within 10 minutes after completion of a standardized breakfast.
  Interventions: Drug: TMC278

INTERVENTIONS:
Drug: TMC278 — 1 25-mg tablet [27.5 mg as the hydrochloride salt) taken orally (by mouth) within 10 minutes after completion of a standardized breakfast on Day 1.

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics and safety of TMC278 after a single oral dose of TMC278 25 mg tablet (27.5 mg as the hydrochloride salt) under fed conditions in healthy Japanese adult male participants.

DETAILED DESCRIPTION:
This is a single center, open-label (all study staff and participants will know the identity of the treatment assigned), single dose study in healthy Japanese adult male participants. The study consists of 3 phases: a screening phase up to 26 days; an inpatient phase from Day -2 to Day 8; and a follow-up assessment phase that occurs on Day 15 (± 2 days) or at the time of the participant's early withdrawal from the study. Participants who meet the selection criteria will be admitted to the investigational institute on two days before the dose (Day -2). All enrolled participants will receive orally (by mouth) a single dose of one TMC278 25 mg tablet on Day 1 within 10 minutes after completion of the standardized breakfast. Enrolled participants will remain in the investigational institute for the entire duration of the inpatient phase. Participants will be discharged on Day 8 after the completion of all required assessments. Blood samples for determination of plasma concentrations of TMC278 will be collected over a period of 168 hours (7 days). The maximum study duration for each participant is 45 days, including the screening phase, in-patient period, and follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Japanese healthy men
* body mass index (BMI) between 18.5 and 25.0 kg/m², inclusive and a body weight of not less than 50 kg

Exclusion Criteria:

* History of or current medical illness considered by the investigator to be clinically significant and should exclude the participant or that could interfere with the interpretation of the study results
* Laboratory abnormality of grade 2 or greater (defined by the World Health Organization Adult Toxicity Table) or clinically significant abnormal values as assessed by the investigators
* Clinically significant abnormal physical examination and vital signs at screening as assessed by the investigators
* Use of any prescription or nonprescription medication (including vitamins and herbal supplements), within 14 days before the dose of TMC278 25 mg tablet
* History of clinically significant drug or food allergies, especially known hypersensitivity and/or known allergy to TMC278 or any of the excipients of the formulation

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2013-03; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
plasma TMC278 concentrations | Baseline (predose) up to 168 hours postdose
  Blood samples will be taken at 16 timepoints: Predose, 0.5, 1, 2, 3, 4, 5, 6, 9, 12, 16, 24, 48, 72, 120, and 168 hours postdose.

SECONDARY OUTCOMES:
The number of participants who experience adverse events | Up to 17 days following study drug administration
  As a measure of safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (1):
- Tokyo, Japan

REFERENCES:
- See also: An Open-label, Single-dose Study to Investigate the Pharmacokinetics and Safety of TMC278 after Oral Administration of TMC278 25 mg Tablet under Fed Condition in Healthy Japanese Adult Male Subjects — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=3849&filename=CR101181_CSR.pdf